CLINICAL TRIAL: NCT04740957
Title: Characterising the Natural History of Mucosal Metabolism During Colorectal Anastomotic Healing
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IRAS 246354
Record Dates: First submitted 2021-02-03; First posted 2021-02-05 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Healing of Colorectal Anastomoses

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observational cohort (No Intervention): 100 patients undergoing elective left colonic or rectal resection with a primary anastomosis will be recruited pre-operatively throughout the study period. This study will not affect or delay the intended treatment for study participants.
  Patients will undergo serial endoscopic examination of the anastomosis post-operatively. Blood, urine, stool, and mucosal biopsies will be serially collected.
- Distal limb feeding cohort (Experimental): This interventional arm will demonstrate the safety of re-introducing ileostomy effluent into the downstream (distal) limb of an ileostomy. The preliminary data will enable exploration of the association between microbiome and post-operative function and enable adequate powering of future interventional studies.
  A subgroup of 20 patients undergoing a resection with a covering ileostomy will be recruited to the intervention arm. Complete healing of the colorectal anastomosis will first be confirmed by water-soluble contrast enema 8 weeks post-operatively (this is standard practice). Patients will be taught how to inject the output from the proximal ileostomy limb into the distal limb (this connects to the colon and thus the colorectal anastomosis) daily until the ileostomy closure date.
  Interventions: Other: Distal limb reintroduction of ileostomy effluent

INTERVENTIONS:
Other: Distal limb reintroduction of ileostomy effluent — Patients will undergo water soluble contrast enema to confirm anastomotic healing 8 weeks post operatively as per standard practice at Imperial.
  Patients will be educated in how to reintroduce ileostomy output to the distal (downstream) loop of their ileostomy. They will be asked to reintroduce 50ml of ileostomy output using a conventional long-tipped bladder syringe daily until surgery to close the stoma.
  Arms: Distal limb feeding cohort

SUMMARY:
This pilot study aims to investigate anastomotic healing and its underlying mechanisms at a mucosal level. It is a first-in-human study which will demonstrate the safety of post-operative endoscopic assessment of a colorectal anastomosis and provide preliminary data in order to power future interventional studies.

100 patients undergoing elective left colonic or rectal resection with a primary anastomosis will be recruited pre-operatively throughout the study period. This study will not affect or delay the intended treatment for study participants.

Patients will undergo serial endoscopic examination of the anastomosis post-operatively. Blood, urine, stool, and mucosal biopsies will be serially collected.

A subgroup of 20 patients with a defunctioning ileostomy will be recruited to an interventional arm. This interventional arm will demonstrate the safety of re-introducing ileostomy effluent into the downstream (distal) limb of an ileostomy. The preliminary data will enable exploration of the association between microbiome and post-operative function and enable adequate powering of future interventional studies.

ELIGIBILITY:
Inclusion Criteria:

Patients undergoing elective left sided colonic or rectal resections with primary anastomosis with or without diverting ileostomy.

Exclusion Criteria:

* Inability to communicate in English
* People who lack capacity to consent
* Emergency colorectal resection whilst awaiting elective surgery
* Age <18
* Permanent stoma formation
* People on long term immunosuppressive medication
* People on long term renal replacement therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-05-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Anastomotic healing | 1 year
  Healing of the colorectal anastomosis when assessed endoscopically - with no visible defects in the anastomosis.

SECONDARY OUTCOMES:
Failure of anastomotic healing | 1 year
  Anastomotic leak detected either by radiological imaging (CT scanning) or a direct return to theatre

OTHER OUTCOMES:
Changes in microbial diversity | 1 year
  Changes in microbial abundance and diversity at the anastomosis. The nature of any change is as yet not investigated and unpredictable - this is an observational outcome measure.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College Healthcare NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No